CLINICAL TRIAL: NCT04196244
Title: INtravenous Contrast Computed Tomography Versus Native Computed Tomography in Patients With Acute Abdomen and Impaired Renal functiOn (INCARO) - a Multicentre, Open-label, Randomised Controlled Trial
Brief Title: Intravenous Contrast Computed Tomography Versus Native Computed Tomography in Patients With Acute Abdomen and Impaired Renal Function
Acronym: INCARO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Sallinen, Adj. Prof., Consultant, Clinical researcher, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: INCARO-HYKS
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Acute Abdomen; Radiocontrast Nephropathy
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal or body CT with intravenous contrast (Experimental): Abdominal or body CT with intravenous contrast
  Interventions: Diagnostic Test: Abdominal or body CT with intravenous contrast
- Abdominal or body CT without intravenous contrast (native CT) (Active Comparator): Abdominal or body CT without intravenous contrast (native CT)
  Interventions: Diagnostic Test: Abdominal or body CT without intravenous contrast (native CT)

INTERVENTIONS:
Diagnostic Test: Abdominal or body CT with intravenous contrast — Abdominal or body CT with intravenous contrast
  Arms: Abdominal or body CT with intravenous contrast
Diagnostic Test: Abdominal or body CT without intravenous contrast (native CT) — Abdominal or body CT without intravenous contrast (native CT)
  Arms: Abdominal or body CT without intravenous contrast (native CT)

SUMMARY:
Computer tomography (CT) is the primary imaging option for acute abdominal pain in adults. Intravenous (IV) contrast media is used to improve the CT quality. In patients with impaired renal function, post-contrast acute kidney injury (PC-AKI) has remained a significant concern. Modern retrospective studies have shown no association between worsened baseline renal function and IV-contrast CT. However, no randomised controlled trial has been done to conclude this. The INCARO (INtravenous Contrast computed tomography versus native computed tomography in patients with acute Abdomen and impaired Renal functiOn) trial is a multicentre, open-label, parallel group, superiority, individually randomised controlled trial comparing IV-contrast enhanced CT to native CT in patients with impaired renal function. Patients requiring emergency abdominal or body CT with eGFR 15-45 ml/min/1.73 m2 are included in the study. The primary outcome is a composite outcome of all-cause mortality or renal replacement therapy within 90 days from CT.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring emergency abdominal or body CT with eGFR 15-45 ml/min/1.73 m2

Exclusion Criteria:

* Age less than 18 years
* Pregnancy
* eGFR less than 15 or more than 45 ml/min/1.73 m2
* Renal replacement therapy within 30 days prior enrolment
* CT with IV contrast less than 72 hours prior enrolment
* Suspicion of vascular occlusion, dissection or bleeding (i.e. need for IV-contrast)
* CT needed without IV-contrast to detect or rule out ureteral stone
* IV contrast allergy
* Inability to give written consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 994 (Estimated)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Mortality or renal replacement therapy | Within 90 days from CT
  A composite outcome that combines all-cause mortality or renal replacement therapy (number of patients)

SECONDARY OUTCOMES:
Acute kidney injury (AKI) grade | Within 72 hours after CT
  The most severe acute kidney injury (AKI) grade defined by KDIGO classification on serum creatinine
Any organ failure | 48 hours after CT
  Any organ failure defined by at least 2 SOFA (Sequential Organ Failure Assessment) points excluding central nervous system (number of patients)
Alive and hospital-free | Within 90 days after CT
  Alive and hospital-free (days)
Time from CT to definitive treatment | During hospital stay estimated on average 7 days
  Time from CT to definitive treatment (i.e. surgery, radiological intervention, endoscopy, medication)

OTHER OUTCOMES:
All-cause mortality | 6 months from CT
  All-cause mortality
All-cause mortality | 1 year from CT
  All-cause mortality
All-cause mortality | 5 years from CT
  All-cause mortality
All-cause mortality | 10 years from CT
  All-cause mortality
Renal replacement therapy | 6 months from CT
  Number of patients requiring renal replacement therapy
Renal replacement therapy | 1 year from CT
  Number of patients requiring renal replacement therapy
Renal replacement therapy | 5 years from CT
  Number of patients requiring renal replacement therapy
Renal replacement therapy | 10 years from CT
  Number of patients requiring renal replacement therapy
Renal transplant | 6 months from CT
  Number of patients undegoing renal transplant
Renal transplant | 1 year from CT
  Number of patients undegoing renal transplant
Renal transplant | 5 years from CT
  Number of patients undegoing renal transplant
Renal transplant | 10 years from CT
  Number of patients undegoing renal transplant

CONTACTS AND LOCATIONS:
Locations (3):
- Finland (3):
  - Jorvi hospital, Helsinki University Hospital, Espoo
  - Meilahti hospital, Helsinki University Hospital, Helsinki
  - Hyvinkää hospital, Hyvinkää

IPD SHARING:
Plan to Share IPD: No
Not shared.

REFERENCES:
- [Derived] Raty P, Mentula P, Lampela H, Nykanen T, Helantera I, Haapio M, Lehtimaki T, Skrifvars MB, Vaara ST, Leppaniemi A, Sallinen V. INtravenous Contrast computed tomography versus native computed tomography in patients with acute Abdomen and impaired Renal functiOn (INCARO): a multicentre, open-label, randomised controlled trial - study protocol. BMJ Open. 2020 Oct 6;10(10):e037928. doi: 10.1136/bmjopen-2020-037928. PMID 33028554